CLINICAL TRIAL: NCT06553417
Title: Effectiveness and Tolerability of an Emollient 'Plus' Compared to Urea 10% in Patients With Mild-moderate Atopic Dermatitis
Brief Title: Emollient 'Plus' vs Urea 10% for Mild-Moderate Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: L'Oreal (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2141/112/2/V/2023
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis; skin barrier; moisturizer; bacterial lysate; clinical efficacy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — N,N'-11-bis((1Z,4Z)-7alphaH-germacra-1(10),4-dienyl)urea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The moisturizer codes will be blinded (double-blind) until all study phases are completed. This ensures that the participants, investigators, and outcomes assessors are unaware of which intervention each participant is receiving during the study. This helps to minimize potential bias in the evaluation of the treatment outcomes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aqua posae + microresyl (Experimental): • Participants in this arm will receive the moisturizer formulation containing aqua posae and microresyl.
  Interventions: Other: Aqua posae and microresyl
- 10% Urea (Active Comparator): • Participants in this arm will receive the moisturizer formulation containing 10% urea.
  Interventions: Other: Urea 10%

INTERVENTIONS:
Other: Aqua posae and microresyl — * This intervention involves the use of two topical products:
    * Aqua posae - a moisturizing agent
    * Microresyl - an active ingredient with potential therapeutic effects
  * Subjects in Group A will be instructed to apply these two products (aqua posae and microresyl) twice daily to the upper and lower limbs, including both lesional and non-lesional areas of the skin.
  The use of these interventions will be evaluated over a 12-week period, with assessments of Transepidermal Water Loss (TEWL), skin hydration, skin pH, index scoring of atopic dermatitis (SCORAD), erythema area severity index (EASI), pruritus visual analogue scale (PVAS), quality of life (DLQI), and any adverse effects.
  Arms: Aqua posae + microresyl
Other: Urea 10% — Intervention 2: Urea 10%
  * This intervention involves the use of a 10% urea-based topical moisturizing product.
  * Subjects in Group B will be instructed to apply the 10% urea moisturizer twice daily to the upper and lower limbs, including both lesional and non-lesional areas of the skin.
  The use of these interventions will be evaluated over a 12-week period, with assessments of Transepidermal Water Loss (TEWL), skin hydration, skin pH, index scoring of atopic dermatitis (SCORAD), erythema area severity index (EASI), pruritus visual analogue scale (PVAS), quality of life (DLQI), and any adverse effects.
  Arms: 10% Urea

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and tolerability of an Emollient Aqua Posae + Microesyl compared to urea 10% in patients with mild-moderate atopic dermatitis The main question it aims to answer is:

" To evaluate the effectiveness and tolerability of an Emollient Aqua Posae + Microesyl compared to urea 10% in patients with mild-moderate atopic dermatitis age 18 years and above". Moisturizer application will be performed twice daily, 3 minutes after bathing, with a standardized dose using the Finger Tip Unit (FTU) method.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years
* AD patients who meet the criteria for AD diagnosis according to the Hanifin-Rajka criteria.
* Patients with mild-moderate AD according to the SCORAD index.
* Patients who have AD lesions on the hands and/or feet.
* Patients with good general condition.
* Patients are willing to participate in the study and sign the informed consent.

Exclusion Criteria:

* Pregnant and lactating patients.
* Patients with a history of allergies to ingredients contained in moisturizers
* Patients who clinically have other skin diseases such as psoriasis, seborrheic dermatitis, contact dermatitis or AD with secondary infections that can affect the SCORAD index parameters, skin hydration, skin pH and side effects on the skin area being assessed.
* Patients receiving topical or systemic immunomodulatory and/or immunosuppressant therapy.
* Patients receiving topical and/or systemic antibiotic therapy
* Patients receiving systemic antihistamine therapy (patients who require antihistamines during the study will be recorded on the observation sheet)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
SCORAD (Scoring Atopic Dermatitis) | Through study completion, 12 week
  * The SCORAD is a composite score that evaluates the extent and severity of atopic dermatitis.
  * The SCORAD scale ranges from 0 to 103, with higher scores indicating more severe disease. The ranges of the SCORAD (0-25 for 'mild' disease, and 25-50 for 'moderate' disease, >50 for severe disease)
PVAS (Pruritus Visual Analog Scale) | Through study completion, 12 week
  * The PVAS is a 100 mm visual analog scale that assesses the severity of pruritus (itching) experienced by the patient.
  * The PVAS ranges from 0 (no itch) to 100 (worst imaginable itch).
EASI (Eczema Area and Severity Index) | Through study completion, 12 week
  * The EASI is a tool that measures the extent and severity of atopic dermatitis lesions.
  * The EASI score ranges from 0 to 72, with higher scores indicating more severe disease. 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe
DLQI (Dermatology Life Quality Index) | Through study completion, 12 week
  * The DLQI is a questionnaire that assesses the impact of skin diseases on a patient's quality of life.
  * The DLQI score ranges from 0 to 30, with higher scores indicating a greater impairment of quality of life.

SECONDARY OUTCOMES:
Transepidermal Water Loss (TEWL) | Through study completion, 12 week
  * TEWL is a measure of the barrier function of the skin, with higher values indicating a more compromised skin barrier.
  * TEWL is typically measured in g/m^2/h.
Skin Hydration | Through study completion, 12 week
  * Skin hydration is a measure of the moisture content of the skin, with higher values indicating more hydrated skin.
  * Skin hydration is typically measured using corneometry, with the values reported in arbitrary units (a.u.).
Skin pH | Through study completion, 12 week
  * Skin pH is a measure of the acidity of the skin surface, with normal skin having a slightly acidic pH around 5.5.
  * Skin pH is measured on a scale from 0 to 14, with lower values indicating more acidic skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kong HH, Oh J, Deming C, Conlan S, Grice EA, Beatson MA, Nomicos E, Polley EC, Komarow HD; NISC Comparative Sequence Program; Murray PR, Turner ML, Segre JA. Temporal shifts in the skin microbiome associated with disease flares and treatment in children with atopic dermatitis. Genome Res. 2012 May;22(5):850-9. doi: 10.1101/gr.131029.111. Epub 2012 Feb 6. PMID 22310478
- [Background] Zelenkova H, Kerob D, Salah S, Demessant-Flavigny AL. Impact of daily use of emollient 'plus' on corticosteroid consumption in patients with atopic dermatitis: An open, randomized controlled study. J Eur Acad Dermatol Venereol. 2023 Jun;37 Suppl 5:27-34. doi: 10.1111/jdv.18947. Epub 2023 Apr 24. PMID 37092256
- [Background] Wollenberg A, Barbarot S, Bieber T, Christen-Zaech S, Deleuran M, Fink-Wagner A, Gieler U, Girolomoni G, Lau S, Muraro A, Czarnecka-Operacz M, Schafer T, Schmid-Grendelmeier P, Simon D, Szalai Z, Szepietowski JC, Taieb A, Torrelo A, Werfel T, Ring J; European Dermatology Forum (EDF), the European Academy of Dermatology and Venereology (EADV), the European Academy of Allergy and Clinical Immunology (EAACI), the European Task Force on Atopic Dermatitis (ETFAD), European Federation of Allergy and Airways Diseases Patients' Associations (EFA), the European Society for Dermatology and Psychiatry (ESDaP), the European Society of Pediatric Dermatology (ESPD), Global Allergy and Asthma European Network (GA2LEN) and the European Union of Medical Specialists (UEMS). Consensus-based European guidelines for treatment of atopic eczema (atopic dermatitis) in adults and children: part I. J Eur Acad Dermatol Venereol. 2018 May;32(5):657-682. doi: 10.1111/jdv.14891. PMID 29676534
- [Background] Ch'ng CC. Rebalancing of the skin microbiome with an emollient 'plus' for effective management of atopic dermatitis: A mini review. Med J Malaysia. 2024 Mar;79(2):203-205. PMID 38553927
- [Background] Gueniche A, Knaudt B, Schuck E, Volz T, Bastien P, Martin R, Rocken M, Breton L, Biedermann T. Effects of nonpathogenic gram-negative bacterium Vitreoscilla filiformis lysate on atopic dermatitis: a prospective, randomized, double-blind, placebo-controlled clinical study. Br J Dermatol. 2008 Dec;159(6):1357-63. doi: 10.1111/j.1365-2133.2008.08836.x. Epub 2008 Sep 15. PMID 18795916
- [Background] Wollenberg A, Kinberger M, Arents B, Aszodi N, Barbarot S, Bieber T, Brough HA, Pinton PC, Christen-Zaech S, Deleuran M, Dittmann M, Fosse N, Gaspar K, Gerbens LAA, Gieler U, Girolomoni G, Gregoriou S, Mortz CG, Nast A, Nygaard U, Rehbinder EM, Ring J, Rossi M, Roxburgh C, Serra-Baldrich E, Simon D, Szalai ZZ, Szepietowski JC, Torrelo A, Werfel T, Flohr C. First update of the living European guideline (EuroGuiDerm) on atopic eczema. J Eur Acad Dermatol Venereol. 2023 Nov;37(11):e1283-e1287. doi: 10.1111/jdv.19269. Epub 2023 Jul 17. No abstract available. PMID 37328919
- [Background] Seite S, Zelenkova H, Martin R. Clinical efficacy of emollients in atopic dermatitis patients - relationship with the skin microbiota modification. Clin Cosmet Investig Dermatol. 2017 Jan 12;10:25-33. doi: 10.2147/CCID.S121910. eCollection 2017. PMID 28138262
- [Background] Magnolo N, Jaenicke T, Tsianakas A, Czech W, Thaci D, Pinter A, Kerob D, Salah S, Luger TA. Comparison of different skin care regimens in patients with moderate to severe atopic dermatitis receiving systemic treatment: A randomized controlled trial. J Eur Acad Dermatol Venereol. 2023 Jun;37 Suppl 5:18-26. doi: 10.1111/jdv.18949. Epub 2023 Apr 24. PMID 37092275